CLINICAL TRIAL: NCT02670642
Title: On Demand vs Continuous Treatment of Endoscopy Negative Subjects With Gastroesophageal Reflux Disease (GERD) With Esomeprazole 20-mg Once Daily Over a 6 Months Long Term Treatment Phase. An Open, Randomised, Multicenter Study. NEED.
Brief Title: Open, Randomised, Multi-center Study of on Demand Versus Continuous Esomeprazole Treatment in Patient With GERD
Acronym: NEED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612C00004
Record Dates: First submitted 2015-12-11; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- On demand 20 mg esomeprazole (Experimental): On demand treatment with 20-mg esomeprazole once daily when needed
  Interventions: Drug: Esomeprazole
- Continuous 20 mg esomeprazole (Active Comparator): Continuous treatment with 20 mg esomeprazole once daily
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
  Other Names: Nexium

SUMMARY:
The purpose of this study is to compare on demand with continuous treatment of endoscopy negative subjects with gastroesophageal reflux disease (GERD), with esomeprazole 20-mg once daily, with regards to willingness to continue in the study as a result of satisfactory treatment over a six-month long term management period, after initial symptom relief.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggestive of GERD, with heartburn as their predominant symptom (described as a burning feeling, rising from the stomach or lower part of the chest up towards the neck), for longer than 6 months.
* Heartburn occurring for 4 days or more during the last 7 days prior to endoscopy. Or, if PPI treatment has been started within the last 7 days prior to endoscopy, then heartburn occurring for 4 days or more during the last 7 days prior to start of PPI treatment
* Male or female, at least 18 years of age (for Austria, at least 19 years of age)
* Have given written informed consent
* Ability to read and write (literate)
* 7 symptom free (from heartburn) days in the last week prior to randomisation (day of visit not included)

Exclusion Criteria:

* Documented esophageal mucosal break
* History of esophageal, gastric or duodenal surgery, except closure and oversewing of an ulcer
* Chronic or recurrent abdominal pain associated with a chronic or recurrent bowel disturbance and/or bloating, that in the opinion of the investigator is likely to be due to irritable bowel syndrome or two or more of the following criteria:

  * Symptoms relieved by defecation
  * Symptoms associated with change in frequency of stools
  * Symptoms associated with change in form of stools
* Any significant "alarm symptoms" such as unintentional weight loss, haematemesis melaena, jaundice or any other sign indicating serious or malignant disease.
* Subjects with current or historical evidence of the following diseases/conditions

  * Zollinger Ellison syndrome
  * Primary esophageal motility disorder(s) i.e. achalasia, scleroderma, esophageal spasm
  * Complications of GERD such as esophageal stricture, ulcer and/or macroscopic Barrett's metaplasia (longer than 3 centimetres) or significant dysplastic changes in the esophagus
  * Evidence of upper gastrointestinal malignancy at the screening endoscopy
  * Gastric and/or duodenal ulcers within the last 2 years
  * Malabsorption
  * Malignancy, or significant cardiovascular, pulmonary, renal, pancreatic or liver disease as judged by the investigator
  * Unstable diabetes mellitus. Stable diabetes controlled on diet, oral agents or insulin is acceptable
  * Cerebrovascular disease, such as cerebral ischemia, infarction, haemorrhage or embolus
* Subjects using a PPI for more than 10 days in the last 28 days, prior to endoscopy
* Use of PPIs for more than 5 days in the last 7 days prior to endoscopy
* Subjects using daily H2-receptor antagonist, prokinetics recommended in the treatment of reflux symptoms or sucralfate during the 2 weeks prior to endoscopy and between the endoscopy and visit 1 and throughout the study
* Need for continuous concurrent therapy with

  * NSAIDs (including selective COX II antagonists, salicylates (unless<165 mg daily for cardiovascular prophylaxis)
  * anticholinergics
  * prostaglandin analogues
  * phenytoin
  * ketoconazole
  * itraconazole
  * warfarin and other vitamin K antagonists
* Pregnancy or lactation. Women of childbearing potential must maintain effective contraception during the study period as judged by the investigator (for Austria: Women of child-bearing potential may only be included when their pregnancy status is assessed by the investigator prior to entry and then at monthly basis. For South-Africa and Spain:

Women of child-bearing potential may only be included when their pregnancy status is assessed by the investigator prior to endoscopy)

* Use of any other investigational compound 28 days prior to start and during the study
* Requirement of an interpreter (illiterate)
* Alcohol and/or drug abuse or any condition associated with poor compliance, including expected non-co-operation, as judged by the investigator
* Previous participation in this study
* Contra-indications to study drugs, e.g. known or suspected allergy to esomeprazole and any other constituents of the formulation. Known hypersensitivity to substituted benzimidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2001-08; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Difference between the proportion of patients who discontinued on-demand esomeprazole treatment versus continuous esomeprazole treatment due to unsatisfactory treatment as determined by the investigator in consultation with the patient | 6 months
  Compare on demand (taken as needed by the patient to adequately control their reflux disease) with continuous treatment of endoscopy negative subjects with gastroesophageal reflux disease (GERD), with esomeprazole 20-mg once daily, with regards to willingness to continue in the study as a result of satisfactory treatment over a six-month long term management period, after initial symptom relief

SECONDARY OUTCOMES:
Reasons for discontinuation of on-demand or continuous esomeprazole treatment assessed by investigator-completed questionnaire at clinical visits | 6 months
Mean number of esomeprazole tablets taken measured using the Medical Event Monitoring System (MEMS) container (date and time of use recorded) | 6 months
Change from baseline in impact of reflux symptoms on health-related quality of life using pre-specified dimensions of the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire | 6 months
Difference between the proportion of patients reporting treatment satisfaction with on-demand versus continuous esomeprazole treatment assessed by standard patient-completed electronic questionnaire at clinical visits and premature discontinuation | 6 months
Frequency of adverse events and assessment of hematology (hemoglobin, leukocytes, thrombocytes) and clinical chemistry (creatinine, alkaline phosphate, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, total bilirubin) | 6 months
Individual patterns of esomeprazole tablet usage measured using the Medical Event Monitoring System (MEMS) container (date and time of use recorded) | 6 months
Change from baseline in impact of reflux symptoms on health-related quality of life using pre-specified dimensions of the Quality Of Life in Reflux And Dyspepsia (QOLRAD) questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Bayerdörffer, MD, Principal Investigator — University Hospital Carl-Gustav-Carus, Medical Clinic and Policlinic I, Fetscherstr. 74, 01307 Dresden, Germany
Locations (60):
- Austria (6):
  - A.ö.Landeskrankenhaus Feldbach, Feldbach
  - A.ö. Landeskrankenhaus Kittsee, Kittsee
  - Spitalverbund Landeskrankenhaus, Knittelfeld
  - Krankenhaus der Stadt Wien, Vienna
  - Hanusch Hospital, Vienna
  - A.ö. Krankenhaus Zell am See, Zell am See
- France (26):
  - 36 boulevard Gambetta, Alès
  - 84 rue Gustave Colin, Arras
  - 15 rue Michelet, Belfort
  - 30 boulevard du Président John Kennedy, Béziers
  - 10 avenue Villeneuve, Cagnes-sur-Mer
  - 13 rue Roquebillière, Cannes La Bocca
  - 91 rue de Paris, Charenton-le-Pont
  - 62 rue Bonnabaud, Clermont-Ferrand
  - 17 villa du Petit Parc, Créteil
  - 24 quai Saint Maurand, Douai
  - 3 place du Marché Couvert, Dreux
  - Clinique Saint Vincent, Épernay
  - 7 rue Parmentier, Épinal
  - Place du Postillon, Issoire
  - 60 rue Jean Bart, Lille
  - 81 avenue du Teil, Montélimar
  - 9 square de Liège, Nancy
  - 6 avenue du Maréchal Juin, Narbonne
  - 74 avenue Paul Doumer, Paris
  - 45bis rue d.Elbeuf, Rouen
  - 64 boulevard Marcel Sembat, Saint-Denis
  - 31 rue Henri Maréchal, Saint-Priest
  - 201 boulevard Robespierre, Talence
  - 4 rue Berlioz, Vélizy-Villacoublay
  - 20 rue de la Glacière, Vitry-sur-Seine
  - 68 avenue Paul Vaillant Couturier, Vitry-sur-Seine
- Germany (14):
  - Wartburgstraße 19, Berlin
  - Gemeinschaftspraxis, Cologne
  - Genovevastraße 5, Cologne
  - Carl Gustav Carus der Tecnischen Universität, Dresden
  - Finkenstraße 31, Freising
  - Reichenbacher Str. 106 a, Görlitz
  - Frankenwaldklinik, Kronach
  - Buchentorstr. 16, Lienen
  - Hammer Str. 108, Münster
  - Albersloher Weg 455, Münster
  - Am Bahnhof 3, Oelde
  - Rudolf-Breitscheid-Str. 56, Potsdam
  - Musikantenweg 3, Ribnitz
  - Friedensstr. 14, Wolmirstedt
- South Africa (9):
  - Gastroenterology Clinic, G73, Department of Internal Medicine, Universitas Hospital, Bloemfontein
  - Burnside House, Room 1, Cape Town
  - Gastroenterology Clinic, E23, Groote Schuur Hospital Observatory, Cape Town
  - Gastroenterology Clinic, Parorama Medi-Clinic, Cape Town
  - Gastroenterology Unit, Room C78, Tygerberg Hospital, Cape Town
  - Unitas Hospital Lyttleton, Centurion
  - Gastroenterology Clinic, Parklands Medical Centre, Durban
  - Gastroenterology Clinic, Milpark Hospital, Johannesburg
  - Gastroenterology Unit, Chris Hani Baragwanath Hospital, Johannesburg
- Spain (5):
  - Centro Médico Teknon, Barcelona
  - Hospital General de Guadalajara, Guadalajara
  - Hospital Central de Asturias, Oviedo
  - Hospital Clínico Universitario, Santiago de Compostela
  - Hospital Virgen Macarena, Seville

REFERENCES:
- [Derived] Bayerdorffer E, Bigard MA, Weiss W, Mearin F, Rodrigo L, Dominguez Munoz JE, Grundling H, Persson T, Svedberg LE, Keeling N, Eklund S. Randomized, multicenter study: on-demand versus continuous maintenance treatment with esomeprazole in patients with non-erosive gastroesophageal reflux disease. BMC Gastroenterol. 2016 Apr 14;16:48. doi: 10.1186/s12876-016-0448-x. PMID 27080034